CLINICAL TRIAL: NCT06867796
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of TL-001 in Healthy Adult Participants
Brief Title: A Safety and Pharmacokinetics Study of TL-001 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TrueLab Biopharmaceutical Co., Ltd (Industry)
Collaborators: Tigermed Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TL-001-101
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- SAD Cohort 1 (Experimental): 8 participants will receive in a 3:1 ratio of a single dose of SAD Dose Level 1 of TL-001 or placebo.
  Interventions: Drug: TL-001; Drug: Placebo
- SAD Cohort 2 (Experimental): 8 participants will receive in a 3:1 ratio of a single dose of SAD Dose Level 2 of TL-001 or placebo.
  Interventions: Drug: TL-001; Drug: Placebo
- SAD Cohort 3 (Experimental): 8 participants will receive in a 3:1 ratio of a single dose of SAD Dose Level 3 of TL-001 or placebo.
  Interventions: Drug: TL-001; Drug: Placebo
- SAD Cohort 4 (Experimental): 8 participants will receive in a 3:1 ratio of a single dose of SAD Dose Level 4 of TL-001 or placebo.
  Interventions: Drug: TL-001; Drug: Placebo
- MAD Cohort 1 (Experimental): 8 participants will receive in a 3:1 ratio of a multiple doses of MAD Dose Level 1 of TL-001 or placebo.
  Interventions: Drug: TL-001; Drug: Placebo
- MAD Cohort 2 (Experimental): 8 participants will receive in a 3:1 ratio of a multiple doses of MAD Dose Level 2 of TL-001 or placebo.
  Interventions: Drug: TL-001; Drug: Placebo

INTERVENTIONS:
Drug: TL-001 — Intravenously administered
Drug: Placebo — Intravenously administered

SUMMARY:
The goal of this study is to evaluate safety, tolerability, pharmacokinetics (PK)), pharmacodynamics (PD) and immunogenicity of single and multiple ascending dose of TL-001 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age.
* Body mass index (BMI) between 18.0 to 32.0 kg/m2 (inclusive), Body weight ≥ 50 kg for males and ≥ 45 kg for females.
* Able to participate and comply with all study procedures and restrictions, and willing to provide written informed consent to participate in the study.
* Female participants who are not pregnant or breastfeeding and meet at least one of the following conditions:

  1. Not of childbearing potential as described in Section 3.7.
  2. Of childbearing potential and agrees to practice abstinence or use highly effective contraception plus condom use as described in Section 3.7 consistently from 30 days prior to Day 1 to the EOS visit.
  3. Should not donate eggs from Day 1 until the EOS Visit.
* Male participants must use condom if sexually active with females of childbearing potential. The female partner of a male participant who does not meet the definition of postmenopausal or permanently surgically sterile is considered of childbearing potential and is required to use a highly effective method of contraception (see Section 3.7) consistently from 30 days prior to Day 1 until the EOS visit of the male participant. Male participants who are surgically sterilized, performed at least 6 months prior to screening, may be enrolled. Male participants must also agree not to donate sperm from Day 1 until the EOS visit.
* No clinically significant findings as determined by medical history, and by results of physical examination, vital signs, ECG, thyroid ultrasound, and clinical laboratory tests obtained within 35 days prior to study treatment administration.

Exclusion Criteria:

* History or presence of any clinically significant organ system disease that could interfere with the objectives of the study or the safety of the participants.
* History of immunological abnormality (i.e., primary or secondary immune suppression) that could interfere with the objectives of the study or the safety of the participants.
* Participants with a significant finding on history of thyroid conditions, thyroid function testing, thyroid antibody testing, or thyroid ultrasound giving reasonable suspicion of a condition that might interfere with the conduct or interpretation of the study.
* Presence or history of any abnormality or illness, which in the opinion of the investigator (or designee) may affect absorption, distribution, metabolism or elimination of the study treatment.
* Any screening laboratory evaluation outside the laboratory reference range that is judged by the investigator (or designee) to be clinically significant, including but not limited:

  1. Participants with eGFR < 80 mL/min/1.73m2 as determined by the CKD-EPI 2021 formula, at the Screening or Baseline visits.
  2. Alanine amino transferase (ALT) or aspartate amino transferase (AST) >1.5 times upper limit of normal (ULN), which remains similar upon repeat, at the Screening or Baseline visits.
  3. Total bilirubin > 1.5 × ULN at the Screening or Baseline visits. Total bilirubin > 1.5 × ULN is acceptable if, direct bilirubin < 40%, normal AST/ALT/ALP, and no evidence of hemolysis, according to investigator (or designee) discretion.
  4. White blood cell count < 3,000 cells/mm3 (< 3.0×109/L) or any abnormal evaluations judged clinically significant by the investigator (or designee) at the Screening or Baseline visits.
  5. Abnormal lipase or amylase level that may interfere with the conduct or interpretation of the study according to investigator (or designee) discretion. Note: If the test results meet the above criteria, a repeat test may be performed to determine eligibility.
* Blood pressure and heart rate are outside the ranges 100-140 mmHg systolic, 50-90 mmHg diastolic, heart rate 40-100 beats/min.
* 12-lead ECG with any abnormality judged by the Investigator (or designee) to be clinically significant, or QTcF interval of > 450 msec for men or >470 msec for women.
* Major surgery or major traumatic injury within 3 months of Day 1. Participants must have also fully recovered from any surgery and/or its complications before initiating the study treatment.
* Malignancy or a history of malignancy prior to the Screening Visit (except for non-melanoma cutaneous malignancies which have been fully treated and completed post-treatment follow-up).
* History of or current active tuberculosis (TB) infection; history of latent TB or current latent TB infection as indicated by a positive QuantiFERON-TB test (or equivalent).
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) antibodies at Screening visit as defined below:

  1. HBV: Positive test for hepatitis B surface antigen (HBsAg).
  2. HCV: Positive test for hepatitis C antibody and a positive test for HCV RNA.
  3. HIV: Positive test for HIV antibody.
* Other active infections or history of infections as follows:

  1. Infection requiring treatment with oral antibiotics, antivirals, antiparasitic, antiprotozoals, or antifungals within 14 days before the Baseline (Day 1) Visit.
  2. A serious infection, defined as requiring hospitalization or IV anti-microbial therapy within 2 months prior to the Baseline (Day 1) Visit.
  3. A history of opportunistic, recurrent, or chronic infections at investigator's (or designee's) discretion.
* History of significant allergy to any medication as judged by the investigator (or designee).
* Use of any prescription medication within 14 days prior to D1 or 5 half-lives, whichever is longer; or use of over-the-counter medications or supplements within 7 days prior to D1 (except for contraception, paracetamol and standard dose of multivitamins).
* Participant has used more than 5 cigarettes per day, or equivalent with other nicotine-containing products, in the 3 months prior to Day 1, or is unwilling to avoid nicotine use during confinement periods.
* Participant who consumes on average more than 14 units of alcohol per week in the 6 months prior to Day 1 (1 unit = 10 mg alcohol), or who has a positive alcohol breath test at Screening or Day -1.
* History of excessive or dependent alcohol or drug use or addiction issues in the two years prior to screening, or participants who are positive for drug testing at screening or Day-1 (Repeat testing will be allowed by the investigator (or designee) discretion).
* Receipt of a live vaccine within 2 months prior to the Baseline visit (participants must agree to avoid live vaccination until at least 3 months after last dose of study drug).
* Receipt of an inactivated vaccine such as COVID-19 vaccination or influenza vaccination, within 14 days prior or planning to receive inactivated vaccine within 14 days post study treatment administration.
* Pregnant or lactating women.
* Cannot commit to full participation in all trial procedures.
* Any other circumstances that, in the Investigator (or designee) judgment, may increase the risk associated with the participant's participation in and completion of the study or could preclude the evaluation of the participant's response.
* Known exposure to anti-TL1A or any type of anti-TL1A therapy.
* Participants who have donated blood or lost a significant amount of blood (>400 mL) within 30 days prior to screening, or who plan to donate blood during the study.
* Participants who have receipt of any study drug or participated in any medical device clinical studies within 30 days or 5 half-lives, whichever is longer prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events adverse events (TEAEs) | Up to 337 Days
  Incidence and severity of AEs, including clinical relevant findings from the clinical laboratory tests (hematology, urinalysis, blood chemistry), physical examination, vital signs, 12-lead ECGs.

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Up to 337 Days
  Time at which Cmax is observed after infusion (tmax)
Maximum concentration (Cmax) | Up to 337 Days
  Maximum observed concentration (Cmax) after infusion
Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | Up to 337 Days
  The area under the plasma concentration-time curve from time 0 to the last measurable time-point (AUC0-t).
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | Up to 337 Days
  The area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf).
Terminal half-life (t1/2) | Up to 337 Days
  The time required for the plasma concentration of the drug to decrease by 50% during the terminal elimination phase
Apparent clearance (CL) | Up to 337 Days
  The volume of plasma cleared of drug per unit time
Apparent volume of distribution (Vz) | Up to 337 Days
  The theoretical volume into which a drug distributes in the body.
Terminal elimination rate constant (λz) | Up to 337 Days
  The rate of drug elimination during the terminal phase of the concentration-time curve.
Percentage of AUC0-inf obtained by extrapolation (%AUCex) | Up to 337 Days
  Percentage of the area under the concentration-time curve from time zero to infinity obtained by extrapolation (%AUCex)
Accumulation ratio (Rac) | Up to 337 Days
  The extent of drug accumulation at steady state compared to the first dose.

OTHER OUTCOMES:
Change from baseline in the serum concentration of pre-specified pharmacodynamic biomarker over time | Up to 337 Days
  Change from baseline in the serum concentration of pre-specified pharmacodynamic biomarker over time.
Incidence of anti-drug antibody (ADA) | Up to 337 Days
  The percentage of participants developing ADA.
Titer of anti-drug antibody (ADA) | Up to 337 Days
  Titer will be measured using an ELISA and reported as endpoint dilution.

IPD SHARING:
Plan to Share IPD: No
TrueLab will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.